CLINICAL TRIAL: NCT01377428
Title: A 12-week Treatment, Multicenter, Randomized, Double Blind, Double Dummy, Parallel-group Study to Assess the Efficacy of Indacaterol (150 μg o.d.) in Patients With Chronic Obstructive Pulmonary Disease, Using Formoterol (12 μg b.i.d.) as an Active Control
Brief Title: Efficacy of Indacaterol 150 µg Versus Formoterol
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQAB149BDE03
Record Dates: First submitted 2011-06-17; First posted 2011-06-21 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2012-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Indacaterol; Formoterol
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — indacaterol; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Indacaterol (Experimental): Indacaterol 150 µg once daily (od) via single-dose dry powder inhaler (SDDPI)
  Interventions: Drug: Indacaterol
- Formoterol (Active Comparator): Formoterol 12 µg twice daily (bid) via single-dose dry powder inhaler (SDDPI)
  Interventions: Drug: Formoterol

INTERVENTIONS:
Drug: Indacaterol — Indacaterol 150 µg once daily (od) via single-dose dry powder inhaler (SDDPI)
  Arms: Indacaterol
Drug: Formoterol — Formoterol 12 µg twice daily (bid) via single-dose dry powder inhaler (SDDPI)
  Arms: Formoterol

SUMMARY:
The study will be a 12 week treatment (84 days), parallel group, randomized, double blind, double dummy, study to assess the superiority of indacaterol (150 μg o.d.) versus formoterol (12 μg b.i.d.) in terms of trough forced expiratory volume in 1 second (FEV1).

Patients will be enrolled after giving informed consent and then begin a screening/run-in period for 14 days. Patients will be randomized to one of two treatment groups using an allocation ratio of 1:1 to receive either indacaterol (150 μg o.d.) and placebo to formoterol, or formoterol (12 μg b.i.d.) and placebo to indacaterol for a treatment period of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD (moderate-to-severe as classified by the Global Initiative for Chronic Obstructive Lung Disease (GOLD) Guidelines, 2009) and:

  * Post-bronchodilator FEV1 <80% and ≥40% of the predicted normal value
  * Post-bronchodilator FEV1/FVC (forced vital capacity) <70%
* Smoking history of at least 10 pack-years

Exclusion Criteria:

* Patients who have had a COPD exacerbation in the 6 weeks prior to screening
* Patients who have had a respiratory tract infection within 6 weeks prior to screening
* Patients with concomitant pulmonary disease
* Patients with a history of asthma
* Patients with diabetes Type I or uncontrolled diabetes Type II
* Any patient with lung cancer or a history of lung cancer
* Patients with a history of certain cardiovascular comorbid conditions

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-09; Primary Completion 2012-02 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
24-h post-dose trough forced expiratory volume in 1 second (FEV1) | After 84 days of treatment

SECONDARY OUTCOMES:
24-h post-dose trough inspiratory capacity (IC) | After 84 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals